CLINICAL TRIAL: NCT02068599
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Topically Applied TV-45070 (4% and 8% w/w Ointment) in Patients With Primary Osteoarthritis Affecting a Single Knee
Brief Title: A Study to Evaluate the Safety and Efficacy of Topically Applied TV-45070 (Ointment) in Participants With Primary Osteoarthritis (OA) Affecting a Single Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TV-45070-CNS-20005
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; OA; Arthritis pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — TV-45070

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TV-45070 4% (Experimental): TV-45070 ointment in a 4% strength applied topically twice daily to the target knee during the treatment period from day 1 through day 28.
  Interventions: Drug: TV-45070
- TV-45070 8% (Experimental): TV-45070 ointment in a 8% strength applied topically twice daily to the target knee during the treatment period from day 1 through day 28.
  Interventions: Drug: TV-45070
- Placebo (Placebo Comparator): Placebo ointment applied topically twice daily to the target knee during the treatment period from day 1 through day 28.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TV-45070 — TV-45070 ointment administered twice a day (morning and evening) to target knee. Participants were provided with a laminated instruction sheet including pictures that both described and illustrated how the ointment was to be spread over the entire knee anteriorly, medially, and laterally in a thin layer that fully covered the area. The ointment was gently massaged into the skin.
  Other Names: funapide; XEN402
  Arms: TV-45070 4%; TV-45070 8%
Drug: Placebo — Placebo ointment matching active intervention administered twice a day (morning and evening) to target knee. Participants were provided with a laminated instruction sheet including pictures that both described and illustrated how the ointment was to be spread over the entire knee anteriorly, medially, and laterally in a thin layer that fully covered the area. The ointment was gently massaged into the skin.
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the change from baseline after 4 weeks of topical administration of TV-45070 (4% and 8% ointment) compared with placebo for the relief of symptoms of primary OA affecting a single knee

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 40 and 85 years of age, Patient has primary OA in a single knee (target knee) confirmed by American College of Rheumatology criteria.
* For patients taking non-steroidal anti-inflammatory drugs (NSAIDs) or other analgesics at the time of the screening visit,
* Patient has visual analog scale (VAS) pain scores with acceptable ranges as determined by the investigator during screening
* Except for OA, patient is judged by the investigator to be medically healthy and able to participate in the study.
* Other criteria apply, please contact the investigator for additional information

Exclusion Criteria:

* Patient has secondary or inflammatory arthritis of the knee such as psoriasis, rheumatoid arthritis (RA), gout, other primary bone disease, or acute trauma.
* Patient has symptomatic chondrocalcinosis
* Patient has a history of fibromyalgia.
* Patient has any painful or disabling conditions that in the opinion of the investigator may confound assessment of pain scoring.
* Patient has uncontrolled cardiac, renal, hepatic or other systemic disorders that in the opinion of the investigator may jeopardize the patient.
* Patient has significant edema or skin disorder (including sores, rashes, or ulcers) at the target knee and surrounding area.
* Patient has a history of total or partial knee replacement in either leg.
* Patient had a major reconstructive knee surgery or arthroscopy of the target knee within 6 months before the screening visit.
* Patient is unable or unwilling to discontinue opioid and/or other prescription analgesics for control of OA pain.
* Patient is intolerant to study drug, its excipients, and/or acetaminophen.
* Patient uses any over the counter oral medications such as glucosamine or chondroitin sulfate products, unless the patient has been receiving the medication for ≥3 months at the time of the screening visit and maintains the medication as stable therapy for the duration of the study.
* Other criteria apply, please contact the investigator for additional information

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2015-04-06 (Actual); Study Completion 2015-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, GCO, Theraputic Area Head, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (42):
- United States (42):
  - Teva Investigational Site 12217, Anaheim, California
  - Teva Investigational Site 12244, Anaheim, California
  - Teva Investigational Site 12252, Cerritos, California
  - Teva Investigational Site 13009, Cerritos, California
  - Teva Investigational Site 12233, El Cajon, California
  - Teva Investigational Site 12240, Lomita, California
  - Teva Investigational Site 12251, Sacramento, California
  - Teva Investigational Site 12234, Spring Valley, California
  - Teva Investigational Site 12256, Clearwater, Florida
  - Teva Investigational Site 12241, DeLand, Florida
  - Teva Investigational Site 12246, Eustis, Florida
  - Teva Investigational Site 12231, Fort Myers, Florida
  - Teva Investigational Site 12216, Hialeah, Florida
  - Teva Investigational Site 12230, Jacksonville, Florida
  - Teva Investigational Site 12220, Miami, Florida
  - Teva Investigational Site 12221, Oldsmar, Florida
  - Teva Investigational Site 12226, Orlando, Florida
  - Teva Investigational Site 12237, Orlando, Florida
  - Teva Investigational Site 12255, Ormond Beach, Florida
  - Teva Investigational Site 12225, Plantation, Florida
  - Teva Investigational Site 12229, Sanford, Florida
  - Teva Investigational Site 12235, Tampa, Florida
  - Teva Investigational Site 12253, Atlanta, Georgia
  - Teva Investigational Site 12250, Marietta, Georgia
  - Teva Investigational Site 12243, Evansville, Indiana
  - Teva Investigational Site 12238, Overland Park, Kansas
  - Teva Investigational Site 12218, New Orleans, Louisiana
  - Teva Investigational Site 12245, Watertown, Massachusetts
  - Teva Investigational Site 12228, Bingham Farms, Michigan
  - Teva Investigational Site 12242, Hazelwood, Missouri
  - Teva Investigational Site 12249, St Louis, Missouri
  - Teva Investigational Site 12223, Omaha, Nebraska
  - Teva Investigational Site 12219, New York, New York
  - Teva Investigational Site 12239, Charlotte, North Carolina
  - Teva Investigational Site 12248, Raleigh, North Carolina
  - Teva Investigational Site 12247, Winston-Salem, North Carolina
  - Teva Investigational Site 12254, Winston-Salem, North Carolina
  - Teva Investigational Site 12224, Cincinnati, Ohio
  - Teva Investigational Site 12236, Memphis, Tennessee
  - Teva Investigational Site 12232, Dallas, Texas
  - Teva Investigational Site 12227, Plano, Texas
  - Teva Investigational Site 12222, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 978 patients with primary OA of the knee were screened for enrollment into this study. 389 patients at 41 centers in the US met entry criteria. Of the 589 patients not enrolled, 551 were excluded on the basis of inclusion/exclusion criteria, 25 patients withdrew consent, and 8 patients were lost to follow-up before the baseline visit.
Pre-assignment Details: After stratification by R1150W polymorphism status: - homozygous minor allele (positive, AA), - heterozygous (positive, AG), and - homozygous common allele (negative, GG), participants were randomly assigned by interactive response technology (IRT) to receive treatment in 1 of 3 treatment groups in a 1:1:1 ratio.
Period: Overall Study
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Started | 130 | 129 | 130
Safety Analysis Set | 129 (One participant withdrew before taking any study drug.) | 128 (One participant withdrew before taking any study drug.) | 130
Full Analysis Set | 129 | 128 | 130
Completed | 119 | 119 | 117
Not Completed | 11 | 10 | 13
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 7 | 5
Not completed — Protocol Violation | 4 | 2 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Noncompliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo | Total
Number analyzed (Participants) | 130 | 129 | 130 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.17) | 59.2 (9.52) | 59.0 (9.65) | 59.5 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 75 | 82 | 228
  Male | 59 | 54 | 48 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 25 | 29 | 74
  Not Hispanic or Latino | 110 | 104 | 101 | 315
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race [Count of Participants; unit: Participants]
  White | 88 | 83 | 88 | 259
  Black | 25 | 33 | 33 | 91
  Asian | 14 | 9 | 8 | 31
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Pacific Islander | 0 | 0 | 0 | 0
  Other | 2 | 4 | 1 | 7
R1150W Polymorphism Status [Count of Participants; unit: Participants] — Patients who carry the R1150W polymorphism have a nucleotide containing adenine (A) instead of guanine (G) in the rs6746030 single nucleotide polymorphism in the SCN9A gene. This change causes an arginine to tryptophan amino acid residue change at position 1150 in the alpha subunit of the voltage-gated sodium channel NaV1.7. Those who carry the R1150W polymorphism may be heterozygous (GA) or homozygous (AA) for the minor allele. This R1150W polymorphism in the SCN9A gene may affect pain perception (Reimann et al 2010).
  Participants
    Homozygous minor allele (positive, AA) | 2 | 3 | 1 | 6
    Heterozygous (positive, AG) | 27 | 28 | 26 | 81
    Homozygous common allele (negative, GG) | 101 | 98 | 103 | 302
Weight [Mean (Standard Deviation); unit: kg] | 79.83 (14.119) | 80.87 (13.010) | 80.29 (13.633) | 80.33 (13.568)
Height [Mean (Standard Deviation); unit: cm] | 168.41 (10.835) | 169.06 (9.927) | 167.99 (9.526) | 168.48 (10.095)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.992 (3.0800) | 28.190 (3.0207) | 28.340 (3.2364) | 28.174 (3.1092)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Last 5 Days of Treatment in the Average Evening Pain Intensity In the Target Knee When Walking on a Flat Surface Using a Mixed Model for Repeated Measures (MMRM)
Description: The Western Ontario and McMasters Universities Arthritis Index [WOMAC] is a widely used, validated, patient-reported questionnaire used to assess pain, stiffness, and physical function in patients with OA of the knee. It consists of 24 items separated into 3 domains (pain [5 items], stiffness [2 items], and physical function [17 items]). WOMAC Question 1 is the first question in the pain domain and asks patients to rate their pain in the target knee while walking on a flat surface. The possible score for each item ranges from 0 (no pain) to 100 mm (worst pain). Participants record their response to WOMAC Question 1 in the study diary based on average pain upon walking since the last assessment or over the past 12 hours. Negative change from baseline scores indicate improvement in pain. MMRM includes week, treatment, study center, and treatment by week interaction as fixed factors; baseline average evening WOMAC Question 1 score as a covariate; and patient as a random factor.
Time Frame: Baseline (day -5 to day -1), Last 5 days of treatment (day 24 to day 28)
Population: The full analysis set (FAS) include all patients in the intent to treat (ITT) population who receive at least 1 dose of study drug and have at least 1 post baseline efficacy assessment. Both baseline and treatment values must be available for a participant to be included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 121 | 123 | 120
units on a scale | -20.56 (1.937) | -23.08 (1.923) | -24.82 (1.928)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; LSM = least square mean; Test type: Superiority; p = 0.1213, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 4.26, 95% CI 2-sided [-1.13 to 9.66]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; LSM = least square mean; Test type: Superiority; p = 0.5231, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 1.74, 95% CI 2-sided [-3.62 to 7.11]

2. Secondary Outcome: Change From Baseline to Last 5 Days of Treatment in the Average Daily WOMAC Pain Subscale Score In the Target Knee Using a Mixed Model for Repeated Measures
Description: The five items in the WOMAC Pain Subscale cover pain during walking, using stairs, in bed, sitting or lying, and standing. Daily WOMAC pain subscale score is calculated as the sum of the 5-item pain subscale scores (WOMAC) recorded at evening for a total range of 0 (no pain) to 500 (worst pain on all 5 items). Negative change from baseline scores indicate improvement in pain. MMRM includes week, treatment, study center, and treatment by week interaction as fixed factors; baseline average evening WOMAC scores for the 5-item pain subscale as a covariate; and patient as a random factor.
Time Frame: Baseline (day -5 to day -1), Last 5 days of treatment (day 24 to day 28)
Population: Full analysis set. Both baseline and treatment values must be available for a participant to be included. For pain subscale, if more than 1 item is missing, the subscale total will not be calculated; otherwise the missing value will be replaced by average of the non-missing values in the subscale.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 121 | 123 | 120
units on a scale | -99.67 (9.365) | -108.52 (9.300) | -117.53 (9.329)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; LSM = least square mean; Test type: Superiority; p = 0.1795, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 17.86, 95% CI 2-sided [-8.26 to 43.98]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; LSM = least square mean; Test type: Superiority; p = 0.4956, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 9.00, 95% CI 2-sided [-16.95 to 34.96]

3. Secondary Outcome: Change From Baseline to Last 5 Days of Treatment in the Average Morning Pain Intensity In the Target Knee When Walking on a Flat Surface Using a Mixed Model for Repeated Measures (MMRM)
Description: The Western Ontario and McMasters Universities Arthritis Index [WOMAC] is a widely used, validated, patient-reported questionnaire used to assess pain, stiffness, and physical function in patients with OA of the knee. It consists of 24 items separated into 3 domains (pain [5 items], stiffness [2 items], and physical function [17 items]). The possible score for each item ranges from 0 (no pain) to 100 mm (worst pain). WOMAC Question 1 is the first question in the pain domain and asks patients to rate their pain in the target knee while walking on a flat surface. Participants record their response to WOMAC Question 1 in the study diary based on average pain upon walking since the last assessment or over the past 12 hours. Negative change from baseline scores indicate improvement in pain. MMRM includes week, treatment, study center, and treatment by week interaction as fixed factors; baseline average morning WOMAC Question 1 score as a covariate; and patient as a random factor.
Time Frame: Baseline (day -5 to day -1), Last 5 days of treatment (day 24 to day 28)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 121 | 122 | 120
units on a scale | -19.84 (1.968) | -21.39 (1.955) | -23.45 (1.956)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Test type: Superiority; p = 0.1963, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 3.61, 95% CI 2-sided [-1.87 to 9.08]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Test type: Superiority; p = 0.4584, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 2.06, 95% CI 2-sided [-3.39 to 7.50]

4. Secondary Outcome: Change From Baseline (Randomization Visit) to the Week 4 Visit in the WOMAC Physical Function Subscale Score for the Target Knee Using a Mixed Model for Repeated Measures
Description: The seventeen items in the WOMAC physical function subscale cover stair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties. WOMAC physical function subscale score is calculated as the sum of the 17-item physical function subscale scores (WOMAC) for a total range of 0 (no pain) to 1700 (worst pain on all 17 items). Negative change from baseline scores indicate improvement in pain. MMRM includes week, treatment, study center, and treatment by week interaction as fixed factors; baseline physical function WOMAC scores for the 17-item subscale as a covariate; and patient as a random factor.
Time Frame: Baseline (day 1, predose), Treatment: Week 4 (day 29)
Population: Full analysis set. Both baseline and treatment values must be available for a participant to be included. For physical function subscale, if more than 3 items are missing the subscale total will not be calculated; otherwise the missing value will be replaced by the average of the non-missing values in the subscale.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 120 | 121 | 118
units on a scale | -372.88 (35.169) | -446.79 (34.812) | -396.39 (35.590)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Test type: Superiority; p = 0.6420, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 23.51, 95% CI 2-sided [-75.83 to 122.84]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Test type: Superiority; p = 0.3141, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -50.40, 95% CI 2-sided [-148.72 to 47.92]

5. Secondary Outcome: Change From Baseline (Randomization Visit) to the Week 4 Visit in the WOMAC Stiffness Subscale Score for the Target Knee Using a Mixed Model for Repeated Measures
Description: The two items in the WOMAC stiffness subscale cover stiffness after first waking and later in the day. WOMAC stiffness subscale score is calculated as the sum of the 2-item stiffness subscale scores (WOMAC) for a total range of 0 (no stiffness) to 200 (worst stiffness on both items). Negative change from baseline scores indicate improvement in stiffness. MMRM includes week, treatment, study center, and treatment by week interaction as fixed factors; baseline stiffness WOMAC scores for the 2-item subscale as a covariate; and patient as a random factor.
Time Frame: Baseline (day 1, predose), Treatment: Week 4 (day 29)
Population: Full analysis set. Both baseline and treatment values must be available for a participant to be included. For stiffness subscale, if both items are missing, the subscale total will not be calculated; otherwise the missing value will be replaced with the non-missing one in the subscale.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 120 | 121 | 118
units on a scale | -45.85 (4.414) | -52.49 (4.358) | -49.01 (4.455)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Test type: Superiority; p = 0.6184, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 3.16, 95% CI 2-sided [-9.31 to 15.63]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Test type: Superiority; p = 0.5775, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = -3.48, 95% CI 2-sided [-15.78 to 8.81]

6. Secondary Outcome: Percentage of Participants With a >=30% and a >=50% Response in Average Evening Pain Intensity of WOMAC Question 1 in the Target Knee During the Last 5 Days of Treatment Compared With Baseline
Description: WOMAC Question 1 is the first question in the pain domain and asks patients to rate their pain in the target knee while walking on a flat surface. The possible score for each item ranges from 0 (no pain) to 100 mm (worst pain). Average pain is calculated using a MMRM which includes week, treatment, study center, and treatment by week interaction as fixed factors; baseline average evening WOMAC Question 1 score as a covariate; and patient as a random factor. Responder rate was calculated as 100 * the value of (average WOMAC pain subscale during the last 5 days of treatment [Days 24 to 28]) - average WOMAC pain subscale at baseline [the 5 days prior to randomization])/average WOMAC pain subscale at baseline (the 5 days prior to randomization). Participants with missing responder rates were treated as nonresponders.
Time Frame: Baseline (day -5 to day -1), Last 5 days of treatment (day 24 to day 28)
Measure: Number; unit: percentage of participants
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 121 | 123 | 120
percentage of participants
  >=50% responder rate | 23.3 | 33.6 | 31.5
  <50% responder rate | 70.5 | 62.5 | 60.8
  >=30% responder rate | 45.0 | 43.8 | 46.9
  <30% responder rate | 48.8 | 52.3 | 45.4
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; >=50% responder rate; Test type: Superiority; p = 0.1011, mixed model for repeated measures — 5% level of significance; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.345 to 1.099]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; >=50% responder rate; Test type: Superiority; p = 0.8400, mixed model for repeated measures — 5% level of significance; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.615 to 1.819]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; >=30% responder rate; Test type: Superiority; p = 0.6607, mixed model for repeated measures — 5% level of significance; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.531 to 1.494]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; >=30% responder rate; Test type: Superiority; p = 0.5777, mixed model for repeated measures — 5% level of significance; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.520 to 1.441]

7. Secondary Outcome: Change From Baseline (Randomization Visit) to the Week 4 Visit in the Pain Quality Assessment Scale - Revised (PQAS-R) for the Target Knee Using a Mixed Model for Repeated Measures
Description: PQAS-R is a standardized self-report tool that measures various aspects of a participant's pain. There are 19 questions (question 19 has 2 parts) that ask the participant to rate the various aspects (intensity, sharpness, heat, cold, etc.) of his/her pain over the past week on average on a scale of 0 to 10 (0 = not [aspect] and 10 = the most or worst imaginable [aspect]). PQAS-R score at each visit is the sum of responses for the 19 questions for a total range of 0=no pain to 200=worst imaginable pain in all aspects. Negative change from baseline scores indicate improvement in stiffness. MMRM includes week, treatment, study center, and treatment by week interaction as fixed factors; baseline PQAS-R score for the 19 questions (20 parts) as a covariate; and patient as a random factor.
Time Frame: Baseline (day 1, predose), Treatment: Week 4 (day 29)
Population: Full analysis set. If any of the 19 questions is missing, the PQAS-R total score will not be calculated for a given visit. If the entire questionnaire is not done at a scheduled time point, it will be considered missing and will not be imputed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 120 | 121 | 118
units on a scale | -39.22 (3.489) | -40.65 (3.453) | -43.16 (3.529)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Test type: Superiority; p = 0.4316, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 3.94, 95% CI 2-sided [-5.90 to 13.79]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Test type: Superiority; p = 0.6126, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 2.51, 95% CI 2-sided [-7.24 to 12.26]

8. Secondary Outcome: Participants' Global Assess of Treatment as Measured by the Patient Global Impression of Change (PGIC) at Weeks 2 and 4 Using a Mixed Model for Repeated Measures (MMRM)
Description: PGIC is a standardized self-report tool that measures the change in a participants overall status rating since the start of treatment on 7-point scale. The 7-point scale is defined as: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. The MMRM model includes week, treatment, study center, and treatment by week interaction as the fixed factors and unconstructed variance-covariance structure.
Time Frame: Weeks 2 (day 15), 4 (day 29)
Population: Full analysis set of participants with data at the timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 129 | 128 | 130
units on a scale
  Week 2: number analyzed (Participants) | 125 | 124 | 120
  Week 2 | 2.87 (0.086) | 2.90 (0.086) | 2.86 (0.088)
  Week 4: number analyzed (Participants) | 120 | 121 | 118
  Week 4 | 2.81 (0.096) | 2.66 (0.095) | 2.60 (0.097)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Week 2; Test type: Superiority; p = 0.9208, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.01, 95% CI 2-sided [-0.232 to 0.257]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Week 2; Test type: Superiority; p = 0.7344, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.04, 95% CI 2-sided [-0.200 to 0.284]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; Week 4; Test type: Superiority; p = 0.1199, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.21, 95% CI 2-sided [-0.056 to 0.486]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; Week 4; Test type: Superiority; p = 0.6357, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.06, 95% CI 2-sided [-0.204 to 0.334]

9. Secondary Outcome: Change From Baseline in the Patient Global Assessment (PGA) Scores at Weeks 2 and 4 Using a Mixed Model for Repeated Measures (MMRM)
Description: PGA is a simple self-report tool for measuring the overall way arthritis is affecting the patient at a particular point in time. There is 1 question and the response is provided on a visual analog scale (VAS) from 0 (very poor) to 100 (very good). The question is: Considering all the ways your arthritis affect you, how are you feeling today? Positive change from baseline scores indicate improvement. The MMRM model includes week, treatment, study center, and treatment by week interaction as the fixed factors; baseline PGA score as a covariate and unconstructed variance-covariance structure.
Time Frame: Baseline (day 1, predose), Week 2 (day 15) and Week 4 (day 29)
Population: Full analysis set of participants with data at the timepoints.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 129 | 128 | 130
units on a scale
  Week 2: number analyzed (Participants) | 124 | 123 | 119
  Week 2 | 4.87 (1.819) | 3.51 (1.808) | 2.10 (1.850)
  Week 4: number analyzed (Participants) | 120 | 120 | 117
  Week 4 | 5.44 (1.949) | 6.35 (1.935) | 4.62 (1.973)
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; Week 2; Test type: Superiority; p = 0.2906, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 2.77, 95% CI 2-sided [-2.377 to 7.916]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; Week 2; Test type: Superiority; p = 0.5892, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 1.41, 95% CI 2-sided [-3.707 to 6.518]
Statistical Analysis 3: Comparison: TV-45070 4% vs Placebo; Week 4; Test type: Superiority; p = 0.7699, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 0.82, 95% CI 2-sided [-4.678 to 6.315]
Statistical Analysis 4: Comparison: TV-45070 8% vs Placebo; Week 4; Test type: Superiority; p = 0.5320, mixed model for repeated measures — 5% level of significance; LSM difference from placebo = 1.74, 95% CI 2-sided [-3.721 to 7.193]

10. Secondary Outcome: Percentage of Participants Who Are Responders Per Outcome Measures in Rheumatoid Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Criteria at Week 4
Description: Participants are classified as 'Yes' if the following criteria are met: - >=50% improvement from baseline and an absolute change >=20 on a scale of 1-100 in either the pain or physical function subscale (WOMAC). or 2 of the 3 criteria as below met: - 1) >=20% improvement from baseline and an absolute change >=10 on a scale of 1-100 in the pain subscale (WOMAC); - 2) >=20% improvement from baseline and an absolute change >=10 on a scale of 1-100 in the physical function subscale (WOMAC); - 3) at least a 20% improvement from baseline and an absolute change >=10 on a scale of 1-100 in PGA. Otherwise, 'No' The responder rate per OMERACT-OARSI criteria was analyzed using a generalized estimating equation (GEE) method, where binary variable responder rate (Yes/No) was modeled through logit link function, with treatment, center, week, and treatment*week as explanatory factors. The unstructured working correlation structure was applied.
Time Frame: Week 4 (day 29)
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 129 | 128 | 130
percentage of participants
  Responder - Yes | 47.3 | 59.4 | 51.5
  Responder - No | 46.5 | 36.7 | 40.8
  Missing | 6.2 | 3.9 | 7.7
Statistical Analysis 1: Comparison: TV-45070 4% vs Placebo; For the responder analyses, participants with missing values were deemed non-responders. Analysis performed using a generalized estimating equation (GEE) method where binary variable responder rate (Yes/No) was modeled through logit link function, with treatment, center, week, and treatment*week as explanatory factors. The unstructured working correlation structure was applied; Test type: Superiority; p = 0.5358, generalized estimating equation (GEE) — 5% level of significance; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.501 to 1.433]
Statistical Analysis 2: Comparison: TV-45070 8% vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.1532, generalized estimating equation (GEE) — 5% level of significance; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.870 to 2.423]

11. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: day 1 up to day 57
Population: Safety analysis population. The safety population includes all randomized participants who receive at least one dose of study medication. In this population, treatment was assigned based upon the treatment participants actually receive regardless of the treatment to which they were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
Number analyzed (Participants) | 129 | 128 | 130
Participants
  Any treatment-emergent adverse event | 43 | 37 | 47
  Treatment-related TEAE | 12 | 10 | 20
  Death | 0 | 0 | 0
  Serious TEAE | 1 | 0 | 1
  Withdrawn from treatment due to TEAE | 3 | 2 | 2

ADVERSE EVENTS:
Time Frame: day 1 up to day 57
Arm/Group | TV-45070 4% | TV-45070 8% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/128 | 0/130
Serious Adverse Events (participants affected / at risk) | 1/129 | 0/128 | 1/130
Other Adverse Events (participants affected / at risk) | 6/129 | 6/128 | 9/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV-45070 4% (N=129) | TV-45070 8% (N=128) | Placebo (N=130)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TV-45070 4% (N=129) | TV-45070 8% (N=128) | Placebo (N=130)
Application site exfoliation (General disorders) | 6 (6) | 6 (6) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data